CLINICAL TRIAL: NCT01445743
Title: Immunogenicity and Safety of an Acellular DPT Vaccine in Pregnant Women in Nuevo Leon, Mexico
Brief Title: Immunogenicity and Safety of an Acellular DPT Vaccine During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Jose M. Ramirez-Aranda, Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EN11-009
Record Dates: First submitted 2011-09-23; First posted 2011-10-04 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Pregnancy
Keywords: Tdap Vaccine; Pregnant woman; Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Biological Products; adacel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biological/Vaccine: Tdap Vaccine (Experimental): Biological: Tdap Intervention women will receive a blinded dose of Tdap vaccine (ADACEL)
  Interventions: Biological: Biological/Vaccine: Tdap Vaccine
- Placebo Comparator: Physiologic Saline solution (Placebo Comparator): Administration of Tdap vaccine or placebo as a single 0.5 mL of Saline (0.9% NaCl) solution
  Interventions: Biological: Biological/Vaccine: Tdap Vaccine

INTERVENTIONS:
Biological: Biological/Vaccine: Tdap Vaccine — Biological: Tdap Intervention comprises 104 randomly assigned pregnant women who will receive a blinded dose of Tdap vaccine (ADACEL) containing 2.5 ug of detoxified pertussis toxin (PT), filamentous haemagglutinin 5 ug, 3 ug Pertactina; 5 ug Fimbriae type 2 and 3, (in addition to Tetanus Toxoid (5 Lf) and diphtheria toxoid (2Lf) as a single 0.5 mL intramuscular injection into the deltoid.
  Other Names: ADACEL

SUMMARY:
That is a double-blind randomized trial with parallel control to demonstrate the safety and immunogenicity of acellular Tdap vaccine in pregnant mexican women. The general objective is to determine the safety and immunogenicity of acellular Tdap vaccine.

The experimental group will receive acellular Tdap vaccine and the control group will receive a placebo consisting of saline 0.9% Sodium Chloride solution, randomly assigned, which will be administered by the same route (intramuscular) and at the same dose (0.5 ml) that the vaccine.

DETAILED DESCRIPTION:
Type of Study: Clinical, randomized, double-blind, parallel control study. Study Subjects: Pregnant women of 19-38years of age, gestational age of 12-24 weeks, low risk of obstetric complications (according to the Obstetric Risk Assessment Form), normal anatomic ultrasound performed in the second quarter of pregnancy and residence in Guadalupe, and Juarez cities in Nuevo Leon State.

The experimental group will receive acellular Tdap vaccine and the control group will receive a placebo consisting of saline (0.9% Sodium Chloride) solution, randomly assigned, which will be administered by the same route (intramuscular) and at the same dose (0.5 ml) that the vaccine by trained personnel.

For both groups, 6 blood samples will be taken. Women: Before and at least 4 weeks after the vaccine or placebo were administered, at hospital admission for delivery. Infant: collected at delivery (cord), 2, 4 and 6 months of age.

Immunogenicity will be compared in both groups by measuring the increase of three of the following antigen-specific antibodies: Pertussis toxin (PT), pertactin (PRN),and fimbriae 2 FIM 2).

Safety Assessment: Each pregnant will be observed at 30 minutes, 24 and 48 hours and one month after the application of the vaccine for side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 38 years
* Pregnancy between 22 and 32 weeks of gestation
* Covered by Ministry of Health medical security
* Definitive residency in Guadalupe and Benito Juarez cities
* Pregnancy termination in the study's hospital.
* At low risk for complication as determined by the obstetrical risk assessment form (ORAF)
* Second trimester or later ultrasound with no significant abnormalities
* Intend to be available for follow up visits and phone calls access through 6 months following delivery
* Willing to give written informed consent

Exclusion criteria:

* Serious mental illness. (Schizophrenia, psychosis, major depression).
* Serious underlying medical condition (e.g Degenerative diseases: Diabetes Mellitus,Hypertension and so on.
* Current smoking or use of drugs.
* Receipt of tetanus-diphtheria toxoid immunization within the past 2 years.
* Be considered as a high risk pregnancy for serious obstetrical complication according to the local Obstetrical Risk Assessment Form.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Elevation of specific pertussis antibody levels in children of women who were administered the immunization | 18 months
  Elevation of at least three antibodies against either pertussis toxin (PT), pertactin (PRN), fimbrial proteins (FIM), or filamentous hemagglutinin (FHA).

SECONDARY OUTCOMES:
Non interference of acellular vaccine in children | 18 months
  To demonstrate the acellular pertussis immunization non interference in the effective development of pertussis antibodies in children at 2, 4, and 6 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ramirez, MD; PhD, Principal Investigator — Proffesor of Family Medicine
Locations (1):
- Hospital Regional Materno Infantil de alta especialidad, Secretaria de Salud de Nuevo Leon, Guadalupe, Nuevo León, Mexico